CLINICAL TRIAL: NCT05801887
Title: Extracorporeal Shock Wave Therapy on Osteoblast-Like Cells In- Vitro Study
Acronym: ESWT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Krishnadevaraya College of Dental Sciences & Hospital (Other)
Responsible Party: Principal Investigator, Dr Prabhuji MLV, Clinical Professor, Krishnadevaraya College of Dental Sciences & Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 02_D012_112292
Record Dates: First submitted 2023-02-06; First posted 2023-04-06 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-03

CONDITIONS: Osteosarcoma
Keywords: ESWT; Cell proliferation; Cell viability
MeSH Terms: conditions — Osteosarcoma; Hyperplasia

STUDY DESIGN:
Intervention Model Description: test group - application of shockwave on osteoblast control group - No shockwave on osteoblast
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Shockwave treated group (Experimental): The osteoblast like cells are treated with shockwaves
  Interventions: Device: Extracorporeal shockwave device
- No shockwave group (Placebo Comparator): The osteoblast like cells are not exposed to shockwaves
  Interventions: Device: No ESWT

INTERVENTIONS:
Device: Extracorporeal shockwave device — Extracorporeal shockwave device generates true shock waves which are characterized by a sudden rise in pressure followed by an exponential decay.
  This is different from the commercially available shockwave devices in which they use piezoelectric based mechanisms which generate high frequency waves.
  Other Names: ESWT
  Arms: Shockwave treated group
Device: No ESWT — the osteoblast like cells are not exposed to shockwaves
  Other Names: shockwave
  Arms: No shockwave group

SUMMARY:
The idea of treating different deformities or diseases in the maxillofacial region with Extracorporeal Shockwave Therapy (ESWT) has recently become popular. It has been widely used in medical practice for the management of urolithiasis, cholelithiasis and in haead and neck region for sialolithiasis. The present study 'Extracorporeal Shock Wave Therapy on Osteoblast-Like Cells In-vitro study' will be done to explore and evaluate the effect of shockwaves. Further, Osteoblast-like cells will be assessed for Cell - Cell interaction and Cell Viability. It will be assessed using a scratch assay, Mtt assay and ATP analysis.

DETAILED DESCRIPTION:
Introduction:

Extracorporeal Shockwave Therapy (ESWT) has recently become popular. Shockwave has been widely used in medical practice for the management of urolithiasis, cholelithiasis and in haead and neck region for sialolithiasis.

Aim:

This study 'Extracorporeal Shock Wave Therapy on Osteoblast-Like Cells In-vitro study' will be done to explore and evaluate the effect of shockwaves. Further, Osteoblast-like cells will be assessed for Cell - Cell interaction and Cell Viability.

Methodology:

In this in-vitro study, 20 Osteoblast - like cells will be included. 10 samples to be considered for Control group and the remaining 10 samples considered as Test group. Extracorporeal shockwave will be applied to the Test samples. They will be further analysed using wound scratch assay which is used to assess Cell proliferative rate and scratch closure through live imaging. MTT assay and ATP assay used to determine Cell viability after exposure to shockwaves. The cell migration and cell viability after exposure to shockwaves will determine its effects on osteoblast-like cells.

ELIGIBILITY:
Inclusion Criteria:

* Cell cultures with a confluency of 70%-80%

Exclusion Criteria:

* Contaminated cell cultures

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-10-22 (Actual); Primary Completion 2022-08-17 (Actual); Study Completion 2022-11-06 (Actual)

PRIMARY OUTCOMES:
Scratch assay | 72hours
  cell migration
MTT Assay and ATP analysis | 74hrs
  Cell viability

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. Roxanne, Bengaluru, Karnataka, India